CLINICAL TRIAL: NCT06955104
Title: A Multi-center, Randomized, Double-blind, Parallel, Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0108+C2407 in Patients With Dyslipidemia
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0108+C2407 in Patients With Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JW24302
Record Dates: First submitted 2025-03-17; First posted 2025-05-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: JW0108 + C2407 (Experimental): For 8weeks QD(Quaque Die)
  Interventions: Drug: JW0108 + C2407
- Control Group: JW0108 + C2407 placebo (Active Comparator): For 8weeks QD(Quaque Die)
  Interventions: Drug: JW0108 + C2407 placebo

INTERVENTIONS:
Drug: JW0108 + C2407 — JW0108 + C2407
  Arms: Experimental Group: JW0108 + C2407
Drug: JW0108 + C2407 placebo — JW0108 + C2407 placebo
  Arms: Control Group: JW0108 + C2407 placebo

SUMMARY:
A Multi-center, Randomized, Double-blind, Parallel, Phase Ⅲ Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of JW0108+C2407 in Patients with Dyslipidemia

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of JW0108+C2407 in dyslipidemia patients

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 years old at the time of written informed consent
* Patients with dyslipidemia

Exclusion Criteria:

* Secondary dyslipidemia
* Patient who does not meet the specified TG, LDL-C level

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in LDL-C | Week 8
  Check LDL-C

SECONDARY OUTCOMES:
Efficacy and Safety: Change from baseline in LDL-C (mg/dL) | Week 8
  Check LDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea